CLINICAL TRIAL: NCT00867984
Title: Torsion Optimization to Reduce Symptoms and Improve Outcomes in Non-responders (TORSION). A Randomized Comparison of Torsion-imaging Guided Optimization vs. Usual Settings.
Brief Title: Torsion Optimization to Reduce Symptoms and Improve Outcomes in Non-responders
Acronym: TORSION
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Calgary (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, Dr. Derek Exner, Professor and Canada Research Chair in Cardiovascular Clinical Trials, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7345220000
Record Dates: First submitted 2009-03-20; First posted 2009-03-24 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Heart Failure, Congestive
Keywords: CRT, resynchronization,
MeSH Terms: conditions — Heart Failure; Creatine deficiency, X-linked

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Torsion-guided VV optimization plus AV optimization.
  Interventions: Other: Torsion optimized
- 2 (Active Comparator): AV optimization only.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Torsion optimized — Torsion optimized VV timing plus AV optimization (VTI)
  Arms: 1
Other: Usual Care — AV optimization (VTI) only
  Arms: 2

SUMMARY:
Approximately 40% of resynchronization therapy recipients do not appear to clearly benefit. These patients are termed 'non-responders'. This study will assess whether a heart ultrasound (echo) technique called 'torsion imaging' can be used to increase the likelihood of benefit from resynchronization therapy.

DETAILED DESCRIPTION:
Background: Despite advances in pharmacotherapy, patients with heart failure (HF) are at high risk for death and hospitalization. Over 25% of patients with systolic HF have dyssynchronous ventricular contraction that impairs left ventricular (LV) function and results in HF progression. Cardiac resynchronization therapy (CRT) is designed to synchronize ventricular mechanical activity, improving cardiac output and reducing HF symptoms. As shown in our pilot data, at least 40% of patients do not respond to CRT despite pre-screening for the presence of longitudinal (long axis) mechanical (velocity) dyssynchrony and targeting LV lead placement to the latest site of latest velocity. Methods to improve the rates of response to CRT are required. Torsion imaging guided optimization of CRT timing is a promising approach and will be tested in this study.

Primary hypothesis: Optimization of inter-ventricular (VV) timing, guided by torsion imaging, will increase functional capacity and reduce LV end systolic volume [ESV] in CRT in patients who have not responded after ≥ 6 months. CRT response will be defined by a ≥ 1 functional class improvement and either a ≥ 10% reduction in LV ESV or a ≥ 5% increase in EF at follow-up versus baseline.

Secondary aims: To compare the following in torsion-guided vs usual care patients: a) echo parameters (intra-LV and VV dyssynchrony and torsion, and mitral regurgitation), b) N-terminal BNP levels, and c) generic / disease-specific quality of life.

Methods: Randomized study of patients who have not responded to CRT after ≥ 6 months.

ELIGIBILITY:
Inclusion Criteria:

* non-response to CRT as indicated,
* stable doses of ACE I / ARB and beta-blocker for ≥ 2 months, &
* controlled heart rate if in atrial fibrillation.

Exclusion Criteria:

* inadequate images to assess torsion
* no significant augmentation in torsion with optimization
* unable or unwilling to provide informed consent,
* medical condition other than HF likely to cause death within 6 months,
* cardiac transplant planned,
* myocardial infarction or revascularization since CRT implant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-03; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Improved functional class (≥ 1 class) & remodeling (either ≥ 10% relative reduction in LV ESV or a ≥ 5% absolute increase in LV EF). | Follow up (3-6 months) versus baseline.

SECONDARY OUTCOMES:
dyssynchrony and torsion | Follow-up (3-6 months) vs. baseline
mitral regurgitation | Follow-up (3-6 months) vs. baseline
N-terminal BNP level | Follow-up (3-6 months) vs. baseline
quality of life | Follow-up (3-6 months) vs. baseline

CONTACTS AND LOCATIONS:
Overall Officials: Derek V Exner, MD, MPH, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada